CLINICAL TRIAL: NCT02444845
Title: Prevalence of Anaemia Secondary to Early Stage Chronic Kidney Disease in High Risk Diabetic and/or Hypertensive Population
Brief Title: Study of Anemia in Chronic Kidney Disease (CKD) Among High-Risk Hypertensive and Diabetic Patients in Pakistan
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML27762
Record Dates: First submitted 2015-05-12; First posted 2015-05-15 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Anemia, Diabetes, Kidney Disease, Chronic, Hypertension
MeSH Terms: conditions — Anemia; Diabetes Mellitus; Kidney Diseases; Bronchiolitis Obliterans Syndrome; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Samples will be collected to determine glomerular filtration rate (eGFR) as well as anemia profile.

GROUPS / COHORTS (1):
- Study Population: Hypertensive and diabetic patients who meet eligibility criteria will be enrolled and evaluated for the presence of anemia secondary to CKD. The first visit will capture medical history including risk factors for CKD; laboratory assessments will be performed at the second and third visits to evaluate glomerular filtration rate (eGFR) and anemia profile, respectively. Participants who are not diagnosted with CKD based upon the second visit will not return for the third visit.

SUMMARY:
The purpose of this study is to evaluate the prevalence of CKD-related anemia at an early stage through screening of high-risk patients in Pakistan at the level of physicians, cardiologists, and diabetologists. The information gathered may serve as a foundation in formulating national guidelines for better early diagnosis and management of patients with CKD.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 40 years
* Known hypertension and/or diabetes for at least 3 years
* Positive dipstick test result for proteinuria

Exclusion Criteria:

* Known CKD
* Receiving erythropoietin
* Blood transfusion within 8 weeks
* History of acute or chronic bleeding, hemolysis, or hemoglobinopathy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll high-risk hypertensive and/or diabetic patients in Pakistan who meet eligibility criteria for observation.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2011-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with anemia secondary to CKD | Up to 12 months

SECONDARY OUTCOMES:
Use of treatment modalities for the management of anemia secondary to CKD | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Pakistan (3):
  - Islamabad
  - Karachi
  - Lahore